CLINICAL TRIAL: NCT00293579
Title: A Phase II Study of Pemetrexed Chemotherapy in Poor-Risk Patients With Advanced Head and Neck Cancer
Brief Title: Pemetrexed Chemotherapy in Poor-Risk Patients With Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-0482
Record Dates: First submitted 2006-02-15; First posted 2006-02-17 (Estimated); Results first posted 2016-03-10 (Estimated); Last update posted 2020-02-10 (Actual); Status verified 2020-01

CONDITIONS: Head and Neck Cancer
Keywords: head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pemetrexed (Experimental): pemetrexed 500 mg/m2 administered iv, every three weeks, for 6 cycles
  Interventions: Drug: Pemetrexed

INTERVENTIONS:
Drug: Pemetrexed — 500 mg/m2 IV every 3 weeks for 6 cycles
  Other Names: ALIMTA

SUMMARY:
This study will estimate overall response rate of pemetrexed in poor risk patients with advanced, metastatic, or recurrent squamous cell carcinoma of the head and neck.

DETAILED DESCRIPTION:
Rationale: Patients with advanced stage head and neck cancer, especially those with disease in the hypopharynx, oropharynx, or oral cavity, and poor performance status defined through clinical testing, are often not eligible for clinical trials and treated with best supportive care. The possibility of developing a well-tolerated chemotherapy regimen in these patients may lead to an equivalent benefit and better palliation. The current study offers the chemotherapy drug pemetrexed to patients with advanced head and neck cancer. Researchers consider this agent to have some anti-tumor efficacy against a variety of site-specific cancers, including head and neck cancer with a response rate that is similar to other single chemotherapy drugs. In addition, previous research indicates that toxicities associated with pemetrexed have been reduced when patients are given folic acid and B12 vitamin supplementation. Along with pemetrexed, the current study provides study participants with both folic acid and B12.

Purpose: The primary objective of this study is to evaluate tumor response, including complete and partial remission, and toxicities from pemetrexed in patients with advanced head and neck cancer. Secondary objectives of this study include measurements of time to tumor progression, survival, and patient quality of life.

Treatment: Study participants will be given pemetrexed through intravenous infusions. Pemetrexed will be administered once every three weeks. This schedule of pemetrexed once every three weeks will be repeated up to six times. Study participants will also be provided with both folic acid and B12 vitamin supplementation before, during, and after study treatments with pemetrexed. Vitamin supplementation is considered critical and compliance must be followed closely. Several tests and exams will be given throughout the study to monitor patients. Treatments will be discontinued due to disease growth and unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Advanced, metastatic, or recurrent head and neck cancers
* Poor risk patients with ECOG performance status of 2

Exclusion Criteria:

* Prior treatment for recurrent or metastatic disease
* No clinical or radiological evidence of brain metatases
* Patients with bone only disease are not eligible
* Patients with pleural or peritoneal effusion as only manifestation of diesase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-02 (Actual); Primary Completion 2008-05 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anterpreet Neki, M.D., Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Derived] Urba S, van Herpen CM, Sahoo TP, Shin DM, Licitra L, Mezei K, Reuter C, Hitt R, Russo F, Chang SC, Hossain AM, Frimodt-Moller B, Koustenis A, Hong RL. Pemetrexed in combination with cisplatin versus cisplatin monotherapy in patients with recurrent or metastatic head and neck cancer: final results of a randomized, double-blind, placebo-controlled, phase 3 study. Cancer. 2012 Oct 1;118(19):4694-705. doi: 10.1002/cncr.27449. Epub 2012 Mar 20. PMID 22434360
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled to the study from March 2006 to January 2008
Period: Overall Study
Arm/Group | Pemetrexed
Started | 5
Completed | 4
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pemetrexed
Number analyzed (Participants) | 5
Age, Continuous [Median (Full Range); unit: years] | 52 [49 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 3 years
Measure: Number; unit: patients
Arm/Group | Pemetrexed
Number analyzed (Participants) | 4
patients | 0

2. Secondary Outcome: Toxicities of Pemetrexed,in Poor Risk Cases With Poor Performance Status and Advanced, Metastatic, or Recurrent Head and Neck Cancer
Description: Drug induced toxicities were assessed and graded according to the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.
Time Frame: Up to 3 years
Measure: Number; unit: percent of patients
Arm/Group | Pemetrexed
Number analyzed (Participants) | 5
percent of patients
  fatigue | 80
  Hypercalcemia | 20
  Anemia | 20

3. Secondary Outcome: Impact of Pemetrexed Chemotherapy on Quality of Life
Description: Quality of life assessements conducted at BL (baseline assessment) and EoT (End of treatment). University of Washington QOL (UW-QOL) questionnaire tests 9 specific areas relating to head and neck cancer. A composite score is calculated by adding together the 9 domain scores to give a scale from 0 (for poor health) to 900 (good health).
Time Frame: Baseline, End of Treatment [up to 3 years]
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pemetrexed
Number analyzed (Participants) | 5
Units on a scale
  Baseline score | 524 (141.6)
  End of Treatment score | 335.5 (185.9)

4. Secondary Outcome: Overall Survival
Description: Overall survival was measured from the time of initial study entry to death due to any cause.
Time Frame: Up to 2 years
Population: All patients were deceased at the time of terminating this study.
Measure: Median (Full Range); unit: months
Arm/Group | Pemetrexed
Number analyzed (Participants) | 4
months | 4.4 [1.4 to 15.4]

ADVERSE EVENTS:
Arm/Group | Pemetrexed
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed (N=5)
Nausea (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 5 (5)
Headache (Nervous system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Increased/Thicker saliva (Gastrointestinal disorders) | 2 (2)
Body jerking (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Gum pain (Gastrointestinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Stomach Pain (Gastrointestinal disorders) | 1 (1)
Loss of balance (Musculoskeletal and connective tissue disorders) | 1 (1)
Increased secretions (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Increased urination (Renal and urinary disorders) | 1 (1)
Vocal changes (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1)
Disorientation (Nervous system disorders) | 1 (1)
Rapid Heart rate (Cardiac disorders) | 1 (1)
Bleeding from Tumor (Vascular disorders) | 1 (1)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alkaline phosphatase (Investigations) | 1 (1)
ALT (Investigations) | 1 (1)
AST (Investigations) | 1 (1)
Gamma-Glutamyl transpeptidase (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes